CLINICAL TRIAL: NCT05735834
Title: Phase 3, Interventional, Multicentre, Open-label, Randomized Study Comparing Rituximab Plus Zanubrutinib to Rituximab Monotherapy in Previously Untreated, Symptomatic Splenic Marginal Zone Lymphoma (RITZ)
Brief Title: Comparison Between Rituximab Plus Zanubrutinib Versus Rituximab Monotherapy in Untreated SMZL Patients
Acronym: RITZ
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IELSG48; 2023-503755-10-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Splenic Marginal Zone Lymphoma
MeSH Terms: interventions — Rituximab; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A - Rituximab + Zanubrutinib (Experimental): Zanubrutinib (160 mg BID orally continuous dosing) is administered for 12 cycles of 28 days each. After cycle 12:
  1. Patients in Complete Response (CR) will stop treatment and enter the follow-up phase.
  2. Patients in partial response (PR) will continue zanubrutinib treatment (160 mg BID orally continuous dosing) for 12 additional cycles of 28 days each for a total of 24 cycles.
  3. Patients in stable disease (SD) or progressive disease (PD) will stop treatment and will enter the follow-up phase.
  Rituximab is infused at the dose of 375 mg/m2 iv on days 1, 8, 15, and 22 of cycle 1 (28 days per cycle), then on day 1 of cycles 3, 6, 9, and 12 (28 days per cycle). After cycle 12:
  1. Patients in CR will stop treatment and enter the follow-up phase.
  2. Patients in PR will go on with rituximab 375 mg/m2 IV on day 1 of cycles 15, 18, 21, and 24 (28 days per cycle).
  3. Patients in SD or PD will discontinue treatment and will enter the follow-up phase.
  Interventions: Drug: Rituximab; Drug: Zanubrutinib
- Arm B - Rituximab (Active Comparator): Rituximab is infused at the dose of 375 mg/m2 iv on days 1, 8, 15, and 22 of cycle 1 (28 days per cycle), then on day 1 of cycles 3, 6, 9, and 12 (28 days per cycle). After cycle 12:
  1. Patients in CR will stop treatment and enter the follow-up phase.
  2. Patients in PR will go on with rituximab 375 mg/m2 iv on day 1 of cycles 15, 18, 21, and 24 (28 days per cycle).
  3. Patients in SD or PD will discontinue treatment and will enter the follow-up phase
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Truxima concentrate for solution for infusion 500 mg/50 ml
  Other Names: Truxima
Drug: Zanubrutinib — Zanubrutinib 80 mg hard capsules
  Other Names: Brukinsa
  Arms: Arm A - Rituximab + Zanubrutinib

SUMMARY:
The goal of this clinical trial is to compare the efficacy and tolerability of the combination of two medicinal products, rituximab, and zanubrutinib, compared to rituximab monotherapy in patients with Splenic Marginal Zone Lymphoma (SMZL), previously untreated and who need systemic treatment.

The main questions it aims to answer are:

* Is the combination rituximab and zanubrutinib a more effective therapy than rituximab monotherapy?
* Is the combination therapy, rituximab and zanubrutinib, well tolerated?

Study participants will be put into one of the two treatment groups (rituximab and zanubrutinib or rituximab alone) for a maximum of two years and will undergo regular visits until three years from treatment start.

DETAILED DESCRIPTION:
Phase III, interventional, multicenter, open label, randomized study to evaluate whether treatment with zanubrutinib in combination with rituximab will result in an improvement in Progression Free Survival (PFS) compared to treatment with rituximab in patients with previously untreated splenic marginal zone lymphoma (SMZL).

Approximately 120 subjects will be randomized in a 1:1 ratio to receive zanubrutinib and rituximab (Treatment Arm A) or rituximab (Treatment Arm B). The study will include a Screening Phase, a Treatment Phase, and a Follow-Up Phase.

Subjects with investigator-confirmed progressive disease (PD) according to the Lugano 2014 criteria or unacceptable toxicity, or investigator/subject decision must discontinue study treatment.

Patients who complete the treatment and patients who will discontinue treatment for any reason will enter the Follow-up Phase.

The Response Follow-up Phase will occur for subjects who complete the treatment or discontinue for reasons other than disease progression and will include efficacy assessments every 24 weeks until investigator-assessed disease progression.

Subjects with PD during the Response Follow-up Phase will continue to be followed in the Survival Follow-up Phase.

An Independent Data Monitoring Committee (IDMC) will be responsible for independent review of the interim safety analysis on the first 20 enrolled patients in the experimental arm.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent in accordance with ICH/GCP regulations before registration and prior to any trial-specific procedures.
* Confirmed diagnosis of SMZL, including Matutes immunophenotype score <3. Evaluation of the following features is desirable: absence of CD103 expression by flow cytometry, absence of Cyclin D1, BCL6, and CD10 expression by immunohistochemistry, and absence of the MYD88 L265P mutation. Patients with prominent splenomegaly and involvement of the splenic hilar and/or extra hilar lymph nodes are eligible
* Previously untreated disease. Patients with prior hepatitis C virus (HCV) infection who underwent HCV eradication and have persistent SMZL after 3 months post-eradication can be included.
* Treatment needs according to the ESMO guideline criteria
* Measurable lesions
* Age ≥ 18 years.
* European Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Absolute neutrophil count (ANC) ≥ 1.0 x 109/L, platelet count ≥ 50 x 109/L, Hb > 7.5 g/dl. Values below such thresholds are allowed if attributable to the underlying lymphoma. Transfusions are allowed if clinically indicated during screening.
* Adequate hepatic and renal function and coagulation parameters
* Patient able and willing to swallow trial drugs as whole tablet/capsule

Exclusion Criteria:

* Previous splenectomy.
* Any systemic therapy for SMZL.
* Patients with central nervous system (CNS) involvement.
* Prior malignancy (other than the disease under study) within the past 2 years, except for curatively treated basal or squamous skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score ≤ 6 prostate cancer.
* Clinically significant cardiovascular disease
* History of cerebrovascular accident or intracranial hemorrhage within 6 months before registration and known bleeding disorders (eg, von Willebrand's disease or hemophilia).
* History of confirmed progressive multifocal leukoencephalopathy (PML).
* Concomitant diseases that require anticoagulant therapy with warfarin or phenprocoumon or other vitamin K antagonists and patients treated with dual anti-platelet therapy. Patients being treated with factor Xa inhibitors (eg, rivaroxaban, apixaban, edoxaban), direct thrombin inhibitors (e. dabigatran) low molecular weight heparin (LMWH), or single anti-platelet agents (eg. aspirin, clopidogrel) can be included but must be properly informed about the potential risk of bleeding.
* Malabsorption syndrome or other condition that precludes the enteral route of administration.
* Any uncontrolled active systemic infection requiring intravenous antimicrobial treatment.
* Known human immunodeficiency virus (HIV) infection.
* Active COronaVIrus Disease 19 (COVID-19) infection or non-compliance with the prevailing hygiene measures regarding the COVID-19 pandemic.
* Active chronic hepatitis C or hepatitis B virus infection
* Active, uncontrolled autoimmune phenomenon (autoimmune hemolytic anemia or immune. thrombocytopenia) requiring steroid therapy with > 20 mg daily of prednisone dose or equivalent.
* Known hypersensitivity to trial drugs or any component of the trial drugs.
* Concomitant treatment with strong CYP3A inducers or inhibitors
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and/or would make the patient inappropriate for enrolment into this trial.
* Pregnancy or breastfeeding.
* Concurrent participation in another therapeutic clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2024-05-21 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) rate at 3 years | From the date of randomization to the date of progression or the date of death from any cause until 3 years after randomization
  PFS is defined as the time from the date of randomization until progression (assessed by the investigator per Lugano 2014 criteria) or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Complete remission rates - Lugano 2014 criteria | At 12 and 24 months after treatment start
  Investigator-assessed complete remission rates achieved at 12 and 24 months of treatment, assessed according to the Lugano 2014 criteria
Best response | From date of treatment start until 24 months after treatment start
  Investigator-assessed best response achieved at any time during the treatment period (24 months) assessed according to the Lugano 2014 criteria
Complete remission rates - Matutes criteria | At 12 and 24 months after treatment start
  Investigator-assessed complete remission rates achieved at 12 and 24 months of treatment, assessed according to the Matutes criteria
Best response - Matutes criteria | From date of treatment start until 24 months after treatment start
  Investigator-assessed best response achieved at any time during the treatment period (24 months) assessed according to the Matutes criteria
Time to next anti-lymphoma treatment (TTNT) | From the end of treatment to the start of the next anti-lymphoma therapy until 3 years after randomization
  Investigator-assessed time to next anti-lymphoma treatment (TTNT) according to the Lugano 2014 criteria. TTNT is defined as time from the end of treatment until the start of the next therapy
Duration of response (DoR) | From the time when criteria for response (ie, CR or PR) are met to the first documentation of relapse or progression until 3 years from randomization
  Investigator-assessed DoR according to the Lugano 2014 criteria
Overall Survival (OS) | From the time of randomization until death as a result of any cause until 3 years from randomization
  OS according to the Lugano 2014 criteria. OS is defined as the time from random assignment until death as a result of any cause
Treatment Emergent Adverse Events (AEs) | From the time of ICF signature until 28 days after treatment discontinuation or until resolution of all treatment-related AEs, whichever occurs later, or starting of a new anti-neoplastic treatment up to 3 years from randomization
  Analysis of type and severity of adverse events (AEs) according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Davide Rossi, MD, Study Chair — Oncology Institute of Southern Switzerland - Bellinzona (Switzerland); Emanuele Zucca, MD, Study Chair — International Extranodal Lymphoma Study Group (IELSG) - Bellinzona (Switzerland); Luca Arcaini, MD, Study Chair — Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
Locations (51):
- Medical University of Vienna, Vienna, Austria
- France (5):
  - Institut Bergonié, Bordeaux
  - CHU de Grenoble, Grenoble
  - Hôpital Saint Louis, Paris
  - Hôpital Lyon-Sud, Pierre-Bénite
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy
- Italy (15):
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - IRCCS AOU di Bologna, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - A.O.U. Policlinico G. Rodolico-S. Marco, Catania
  - IRCCS IRST Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori", Meldola
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo
  - IRCCS Policlinico San Matteo, Pavia
  - Ospedale Santa Maria delle Croci, Ravenna
  - USL-IRCCS of Reggio Emilia, Arcispedale Santa Maria Nuova, Reggio Emilia
  - Policlinico Santa Maria alle Scotte, Siena
  - Ospedale di Circolo e Fondazione Macchi - ASST dei Sette Laghi, Varese
- Norway (2):
  - Oslo University Hospital, Oslo
  - St Olavs Hospital, Trondheim
- Spain (15):
  - Hospedal Clinic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Istitut Català d'Oncologia, Hospital Duran i Reynals, Barcelona
  - Hospital Universitario Cruces, Bilbao
  - Hospital Virgen Arrixaca, El Palmar
  - Clinica Universidad de Navarra, Madrid
  - Hospital 12 De Octubre, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital De Salamanca, Salamanca
  - Hospital De Donostia, San Sebastián
  - Hospital Clinico De Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Karolinska University Hospital, Stockholm, Sweden
- Switzerland (2):
  - Oncology Institute of Southern Switzerland, Bellinzona
  - INSELSPITAL, Bern University Hospital, Bern
- United Kingdom (10):
  - University Hospitals Dorset, Bournemouth
  - University Hospital of Wales, Cardiff
  - Hospital Beatson West of Scotland Cancer Centre, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Clatterbridge Cancer Centre, Liverpool
  - University College London Hospitals, London
  - Guy's Hospital - Guy's and St. Thomas' NHS Foundation Trust, London
  - The Christie, Manchester
  - Churchill Hospital, Oxford
  - The Royal Marsden NHS Foundation Trust, Sutton